CLINICAL TRIAL: NCT05716308
Title: The Effect Evaluation of Continuous Nursing Intervention in Patients With Type 2 Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Hui Du, doctor, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BeijingTH001
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Continuous nursing intervention was performed on the basis of the control group
  Interventions: Behavioral: A continuous nursing intervention group was established.
- control group (No Intervention): discharge guidance was performed according to routine nursing intervention at the time of discharge, and the patients were informed to return to the hospital for regular review (review was performed at 1 month, 3 months, half a year, 1 year, and 2 years after discharge, respectively).

INTERVENTIONS:
Behavioral: A continuous nursing intervention group was established. — Intervention group: Continuous nursing intervention was performed on the basis of the control group: ①A continuous nursing intervention group was established. The group members included chief physician, attending physician, head nurse, specialist nurse and nutritionist. ②The establishment of patient records, patients admitted to hospital by the primary nurse to record the basic situation of patients, including name, age, history of diabetes, DR staging, vision and blood glucose before treatment and other information. ③Personalized nursing intervention was given during hospitalization. Systematic health education was carried out for patients on admission. Targeted psychological counseling was given to some patients. ④After discharge to give continuous care, organize patients to join the WeChat group, group to share knowledge of DR-related diseases, to understand the patient 's medication, diet, vision, the patient 's questions and problems to guide and improve.
  Other Names: The establishment of patient records, patients admitted to hospital by the primary nurse to record the basic situation of patients; Personalized nursing intervention was given during hospitalization; After discharge to give continuous care, organize patients to join the WeChat group, group to share knowledge of DR-related diseases
  Arms: intervention group

SUMMARY:
Objective: To evaluate the application effect of continuous nursing intervention in type 2 diabetic retinopathy (DR), and to explore its clinical application value. Methods：Patients with type 2 DR admitted to our Hospital from June 2019 to June 2022 were selected as the research objects and divided into intervention group and control group by random number table method. The control group received routine nursing intervention, and the intervention group received continuous nursing intervention on the basis of the control group. The related effect evaluation indexes such as fasting blood glucose, 2-hour postprandial blood glucose, glycosylated hemoglobin and visual acuity were collected and compared between the two groups at discharge, 1 year and 2 years after discharge. The readmission rate of the two groups was counted to evaluate the effect of continuous nursing intervention.

ELIGIBILITY:
Inclusion Criteria:

* (1) DR diagnosis and classification criteria in line with the latest version of the 2017 Clinical Guidelines for Diabetic Retinopathy developed by the American Eye Association [9];
* (2) Type 2 diabetes course of more than 5 years, with varying degrees of retinopathy;
* (3) Monocular disease, no blindness;
* (4) Education level above primary school; - (5) Patients informed consent for this study and signed a consent form.

Exclusion Criteria:

* (1) with severe cerebral hemorrhage or cerebral infarction, severe nephrotic syndrome, senile dementia, cardiovascular and cerebrovascular diseases;
* (2) Patients with macular edema, severe corneal (and) or lens opacity affect the observation of the fundus, angle-closure glaucoma can not mydriasis, other fundus diseases, and nursing interventions for other chronic diseases. This study was approved by the ethics committee of our hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
DR patient care satisfaction questionnaire during follow-up | 2 years
  Each item was scored according to three levels of 10 points, 6 points and 2 points, with a total score of 20-100 points. The higher the score, the higher the nursing satisfaction
The Summary of Diabetes Self-Care Activities (SDSCA) | 2 years
  The translated Chinese version of the SDSCA scale consists of 11 items, reflecting five parts of self-management : diet, exercise, blood glucose monitoring, foot care, and drugs. Each item is scored by 8 levels of 0-7 points, of which 1 item is a reverse question. The purpose of this scale is to measure the self-management behavior of patients within 7 days. The total score is 0~77 points. The higher the score, the better the self-management ability. Above 56 points is good for self-management ability, 42~56 points is medium, and below 42 points is poor.
Criteria for visual acuity changes | 2 years
  1. Significant improvement: visual acuity improvement≥4 lines.
  2. improvement: vision improvement≥2 lines.
  3. unchanged: visual acuity increased by 1 line or decreased by 1 line.
  4. decline: visual decline≥2 lines.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital,Capital Medical University, Beijing, Beijing Municipality, China